CLINICAL TRIAL: NCT05177692
Title: A Prospective Clinical Trial to Evaluate an Automated Cerebral Ventricular Drainage System in Patients in the Neurointensive Care.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Skane University Hospital (Other)
Responsible Party: Principal Investigator, David Cederberg, Senior Consultant, Chief of Neurointensive Care Unit, Skane University Hospital, Lund, Sweden, Skane University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIV-21-06-036906
Record Dates: First submitted 2021-12-14; First posted 2022-01-04 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: ICP Regulation Using a New Device for Automated Zero-calibration for a Ventricular Drainage System

STUDY DESIGN:
Intervention Model Description: Intervention group will be compared to a control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group - Vguard (Active Comparator): Intervention group will be fitted with a Vguard system Patients will have double ICP monitoring using the intraventricular drainage and and intraparenchymal ICP monitoring device
  Interventions: Device: Vguard
- Control group - regular intra-ventricular drainage (No Intervention): Control group will be fitted with a standard system for drainage of ventricular fluid Patients will have double ICP monitoring using the intraventricular drainage and and intraparenchymal ICP monitoring device

INTERVENTIONS:
Device: Vguard — VGuard is a system that has been created to ensure that the patients´ ventricular drainage system and pressure monitor closely follows the patient when the head is adjusted vertically. The system consists of a pressure sensor that is connected to the patients´ head. The pressure sensor is connected to a motorized column that automatically adjusts to keep the zero level at level with the patients´ head at all times.
  Other Names: Regular system for intraventricular drainage
  Arms: Intervention group - Vguard

SUMMARY:
This is a prospective, randomised trial to evaluate a new medical device for automated zero calibration of ventricular drainage systems in neurointensive care patients.

Patients will be randomised into the medical device group, or a control group with a standard system for ventricular drainage.

All patients will be fitted with an intraparenchymal ICP monitor, and an ICP monitor connected to the ventricular catheter.

Since ICP monitoring using the ventricular catheter system is reliant upon regular zero-calibrations of the system in relation to the mid-point of the patient head, the ICP value from the intraparenchymal ICP monitor will be used as standard, and the intra-ventricular ICP measurements will be compared to this ICP.

The difference in ICP between the two ICP monitors will be the primary outcome for this trial, where the medical device tested is designed to constantly zero-calibrate the ventricular catheter in relation to the patients´ head.

Secondary outcome of this trial will be number of manual zero-calibrations performed, and number of automated zero-calibrations performed by the device, and AE, SAE and DDs.

DETAILED DESCRIPTION:
Introduction

There is a diversity of acute conditions that may affect the brain, many of which need emergent treatment in a neurointensive care unit with a combination of neurosurgery and neurointensive care. Neurosurgery aims at, when possible, remove pathologies that cause increased pressure on the brain, for example tumors, intracerebral hematomas or, in some cases, cerebrospinal fluid. The neurointensive care aims at diminishing the secondary events that may arise as a direct cause of the initial pathology, for example additional bleedings, brain swelling, stroke etc. Many patients that receive neurointensive care, are fitted with a ventricular drainage (V drain) that is surgically implanted into the fluid filled cavities in the center of the brain. The V drain serves to keep the amount of cerebrospinal fluid at normal levels, but is also used to monitor the intracranial pressure (ICP). By draining the cerebrospinal fluid, ICP can usually be kept at close to normal levels. The V drain is connected via a tubing system to a fluid canister to the side of the patient. The canister can be positioned at different levels in relation to the patient´s brain, allowing for drainage of cerebrospinal fluid when the ICP reaches a certain level. In order to define the so called "zero level", i.e. the level from which the ICP is measured, and the level from which the canister is raised in order to define at which pressure the cerebrospinal fluid should start to drain, a laser pointer is usually directed at the level of the patient ear. In patients that are nursed on the side, the pointer is directed at a point between the eyes, or in the middle of the skull.

Each time a patient is moved, the "zero point" must also be corrected in order for the ICP measurements to be correct, and to make sure that the patient does not over- or under drain cerebrospinal fluid. In a patient that is in a medical coma, this may occur 6-12 times during 24 hours, whereas in an awake patient, it may occur several times an hour.

If the patient´s head suddenly would be high above the zero point, such as when a patient goes from supine to sitting position, the V drain may drain the ventricular system for cerebrospinal fluid quite rapidly. This may result in bleedings on the exterior of the brain due to the collapsed ventricular system, and the patient will get severe headache as a result of the greatly decreased ICP. If the patient´s head is far below the zero level, underdrainage and increased ICP with headache and, in worst case coma may result.

Vguard is a system that has been created to ensure that the patients´ ventricular drainage system and pressure monitor closely follows the patient when the head is adjusted vertically. The system consists of a pressure sensor that is connected to the patients´ head. The pressure sensor is connected to a motorized column that automatically adjusts to keep the zero level at level with the patients´ head at all times. The idea for the system came from an employee at the neurointensive care unit (NICU) at Skane University Hospital, Lund and was developed in collaboration with the regional innovation company, Innovation Skåne.

The investigators have chosen to perform a clinical trial with Vguard, in order to assess its reliability in a clinical environment.

Study Objectives The primary objective of this study is to evaluate the Vguard systems´ ability to automatically zero level a ventricular drainage system compared to patients without the Vguard system.

The secondary objectives of this study are to evaluate safety of the Vguard system in a clinical environment and its´accuracy compared to manual zero levelling each time the patient is moved and a manual zero levelling would take place. In addition, we will measure the number of zero levelings that are initiated automatically by the system, at times when the nursing staff would not deem zero leveling necessary.

Study Plan and Procedures

The study is prospective, randomized and interventional.

Primary outcome for this study will be the difference in mm Hg between intraventricular ICP measured via the V drain and an intra-parenchymal ICP monitor over the duration of the study time.

Secondary outcomes will be number of AE and SAE registered with the Vguard system, the difference in mm Hg between the manual zero level and automated zero level measured at every point that manual zero leveling is performed and the number of automated zero level settings where manual zero leveling has not been deemed necessary by the nursing staff.

Primary end point for this study aims to compare the Vguard systems´ability to regulate ICP with the normal system for ventricular drainage.

Secondary end points for this study aims to evalutate safety of the Vguard system by measuring the number of AE and SAE´s that occur during the course of the trial. The second secondary end point aims to measure the Vguard systems´ability for automated zero-calibration in comparison to manual zero-calibration, and the sensibility of the system for automated zero-calibration, when the nursing staff did not notice a need for it.

Patients that fit the inclusion criteria will be asked to participate via next of kin when admitted to the NICU at Skane University Hospital, Lund. If consent is given, the patient will be enrolled in the study. After enrolment in the study, randomization will take place and the patient will either be fitted with a Vguard system or not. ICP from the V drain and the intra-parenchymal ICP monitor will be recorded during the entire time period during which the patient needs a V drain. Each time the patient is moved or moves, and manual zero leveling is deemed necessary, the nursing staff will perform manual zero leveling and note the difference between the automated and the manual zero leveling. A logging device will be connected to the Vguard system for later comparison between the number of manual adjustments and the number of actual, automated adjustments.

Study duration Each patient will be included in the study for the duration of the time they need a V drain. (Usually 7-14 days) The study is anticipated to run for a time period no longer than 18 months.

Patient monitoring - upon arrival at NICU Patients will be treated and monitored according to standard treatment algorithms based on the underlying pathology.

Extra monitoring device for the study Each patient that is included in this study, will be fitted with a Moberg Component Neuro monitoring System (CNS) that will allow for high resolution data sampling of ICP measured from the V drain and the intra-parenchymal ICP monitor.

V drain manual zero level Patient zero level will be performed according to protocol. Each time the nursing staff plans for a zero leveling, date and time is noted in the research form. (Appendix A) Zero leveling is performed according to local routines, using a laser pointer with a spirit level. If there is a difference between the auto zero leveling already performed by the Vguard system, this difference is measured using a ruler with a mm Hg scale and noted in the research form.

V drain automated zero level Each time the Vguard system performs an automated zero leveling, this is noted in the attached logging device for later comparison between the manual zero leveling and the possible automated zero levels that may occur when the zero level of the patient is slightly off, but not enough for the nursing staff to notice it.

Study Measurements and Endpoints

In this study the following data will be measured/recorded.

Physiological and clinical data Age, gender and primary diagnosis at admission will be noted in the CRF. Patient ICP, measured via the automatically zero leveled system and via the intra-parenchymal ICP monitor will be recorded continuously.

V drain open or closed The patency of the V drain as a reliable ICP measuring device depends on it being closed. If the patient V drain is open for drainage of cerebrospinal fluid, it will be closed hourly for 5 minutes, in order for it to give a reliable ICP measurement to compare with the intra-parenchymal ICP monitor readings. Closure of the V drain will be noted on the Moberg monitor.

Primary end point Mean difference in ICP measured from the closed V drain compared with ICP, measured by the intra-parenchymal ICP monitor.

Secondary end points Mean difference in mm Hg after manual zero leveling compared to the automated zero leveling.

Number of automated zero leveling counts compared to number of manual zero leveling counts.

Monitoring of the trial The trial will be monitored by an independent and certified monitoring body to ensure that the trial is conducted according to good clinical practice SS-EN ISO 14155:2020.

Statistical Methods

ICP measured with V drain vs. intra-parenchymal ICP monitor

The difference between ICP measured with V drain vs. intra-parenchymal ICP monitor at every measuring point will be compared between the interventional and control group using students t-test.

Mean difference in mm Hg is estimated to be 5 +/- 2 in control group Mean difference in mm Hg is estimated to be 2 in interventional group

Power to reach statistical significance of p less than 0,05 = 14 patients in each group

Distance in mm between manual zero point, measured by laser and automated zero point adjusted by Vguard - interventional group only

Will be presented as a mean value per participant and for the group.

Number of automated zero adjustments by Vguard vs. number of manual zero adjustments - interventional group only

No statistical analysis will be performed. Data is presented as numbers.

Publication policy All results of this investigation will be submitted for publication in an appropriate peer-reviewed scientific journal within 3 months after termination of the investigation. All anonymized data will be available at request for a time frame of 10 years, after which these records will be destroyed.

ELIGIBILITY:
Inclusion Criteria:

* Adult of either gender between 18 and 80 years
* Requiring treatment at the NICU for a pathology that needs a V drain combined with an intra-parenchymal ICP monitor.

Exclusion Criteria:

• Withdrawal from study based the will of next of kin or patient

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-12-29 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-03-12 (Actual)

PRIMARY OUTCOMES:
Mean difference in mm Hg between intraventricular ICP measured via the V drain and an intra-parenchymal ICP monitor over the duration of the study time. | 5-21 days
  All patients will be fitted with two ICP monitors, of which one will be the intraventricular drainage, which is dependent upon continuous zero calibration of the pressure dome in relation to the patients head.

SECONDARY OUTCOMES:
Number of AE and SAE registered with the VGuard system | 5-21 days
  AE and SAE specified in Clinical Study Protocol
Difference in mm Hg between the manual zero level and automated zero level measured at every point that manual zero leveling is performed | 5-21 days
Number of automated zero level settings where manual zero leveling has not been deemed necessary by the nursing staff. | 5-21 days

CONTACTS AND LOCATIONS:
Overall Officials: Niklas Marklund, Professor, Principal Investigator — Professor of Neurosurgery
Locations (1):
- Dept of Neurosurgery, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No
The data collected will be handled in a pseudonymized order. The only data from the participants medical records that will be used in this study is demographic data (age/date of birth, gender and diagnosis at inclusion.